CLINICAL TRIAL: NCT04681079
Title: A 2-Period, Crossover Study to Assess the Impact of Nebulizer With Filtered Mouthpiece vs MDI With Spacer on Viral Load in Rooms of Subjects With Mild to Moderate COVID-19
Brief Title: Comparison of Viral Particle Dispersion Following Administration of an MDI or Nebulizer in Subjects With COVID-19
Status: Completed | Type: Observational
Sponsor: Theravance Biopharma (Industry)
Responsible Party: Sponsor
Other Study IDs: 0192
Record Dates: First submitted 2020-12-22; First posted 2020-12-23 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: COVID-19
Keywords: Nebulizer; MDI; Meter Dosed Inhaler; Filter; Spacer; COVID-19; Coronavirus disease 2019; SARS-CoV-2; Aerosol; Viral transmission
MeSH Terms: conditions — COVID-19 | interventions — Albuterol; Nebulizers and Vaporizers

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Crossover Sequence 1: Subjects randomized to receive commercially available albuterol sulfate via MDI with spacer first, followed by albuterol sulfate via nebulizer with filtered mouthpiece.
  Interventions: Drug: albuterol sulfate (MDI); Drug: albuterol sulfate (nebulizer)
- Crossover Sequence 2: Subjects randomized to receive commercially available albuterol sulfate via nebulizer with filtered mouthpiece first, followed by albuterol sulfate via MDI with spacer.
  Interventions: Drug: albuterol sulfate (MDI); Drug: albuterol sulfate (nebulizer)

INTERVENTIONS:
Drug: albuterol sulfate (MDI) — albuterol sulfate inhalation aerosol delivered via metered-dose inhaler (MDI) with spacer
Drug: albuterol sulfate (nebulizer) — albuterol sulfate inhalation aerosol delivered via nebulizer with filtered mouthpiece

SUMMARY:
A randomized, 2-period crossover, single-center, open-label study for viral sample collection. After initiation of inhaled therapy with nebulizer or MDI, cascade impactors and surface samplers will be used to assess viral loads in rooms of subjects with COVID-19.

DETAILED DESCRIPTION:
Observational Study Model = Other [non-treatment; impact on external location (rooms and surfaces)]

Time Perspective = Other [viral load samples taken at various time points after nebulization or MDI administered]

Sampling Method = Non-probability sample [to be described by study team]

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent, either themselves or via legally acceptable representative, prior to undergoing study procedures
2. Willing and able to comply with study-related procedures/assessments
3. Adults over 18 years of age
4. COVID-19 infection as confirmed by PCR from nasopharyngeal, oropharyngeal swabs and/or saliva specimen taken within the previous 5 days

Exclusion Criteria:

1. Subjects currently receiving mechanical ventilation or noninvasive positive-pressure ventilation, or subjects who, in the opinion of the investigator, will require ventilatory support (i.e., mechanical ventilation or noninvasive positive-pressure ventilation) within the next 12 hours Note: Signs of impending need for ventilatory support include pronounced hypoxia despite supplemental oxygen >6 L/min, prolonged respiratory rate (i.e., >30 breaths per minute), signs of respiratory muscle fatigue, or paradoxical diaphragm.
2. Presence of significant comorbidity that, in the opinion of the investigator, makes the subject unsuitable for participation in the study
3. Known or suspected hypersensitivity to albuterol, history of paradoxical bronchospasm, or significant cough response to albuterol
4. Participating in other clinical trials related to COVID-19 thought to interfere with study interpretation (e.g., antivirals or antibodies that might change the viral load over the course of a day; subjects should not receive antibody therapy within 24 hours before the baseline period)
5. Active or incompletely treated pulmonary infections, such as tuberculosis (or known history of nontuberculosis mycobacterium) over past 12 months
6. Pregnant or currently breast feeding, or a positive urine pregnancy dip test performed at baseline (women only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with mild to moderate COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2021-05-04 (Actual); Primary Completion 2021-11-22 (Actual); Study Completion 2022-01-18 (Actual)

PRIMARY OUTCOMES:
Viral Load | Baseline, Day 1
  Change in viral load from baseline at each sample point (room air and surfaces). This outcome measure is listed as exploratory in the protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Theravance Biopharma
Locations (1):
- Theravance Biopharma Investigational Site, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No